CLINICAL TRIAL: NCT02716753
Title: The Effects of Male Factors on the Success Rate of in Vitro Fertilization. Will Deposition of Seminal Plasma Around the External Cervical os Increase Pregnancy Rate?
Brief Title: Effects of Seminal Plasma on Pregnancy Rate With IVF
Acronym: SENAVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostergotland County Council, Sweden (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Elizabeth Nedstrand, MD, PhD, Ostergotland County Council, Sweden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dno 2015/387-31
Record Dates: First submitted 2016-03-17; First posted 2016-03-23 (Estimated); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Seeds

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Seminal plasma (Experimental): Half of the amount of seminal plasma received after preparation of the spermatozoa used for IVF will be deposited around the external cervical opening
  Interventions: Biological: seminal plasma
- Physiological NaCL solution (Placebo Comparator): An amount of physiological NaCL solution equal to half of the amount of seminal plasma received after preparation of the spermatozoa used for IVF will be deposited around the external cervical opening
  Interventions: Biological: Physiological NaCL solution

INTERVENTIONS:
Biological: seminal plasma
  Arms: Seminal plasma
Biological: Physiological NaCL solution
  Arms: Physiological NaCL solution

SUMMARY:
All couples planned for IVF will be asked to participate. After information and received informed consent they will be randomized into two groups.

At the time for ovum pick up during an IVF procedure either half of the amount of seminal plasma or the same amount of physiological NaCl solution will be installed around the external cervical opening in vagina. The syringe with seminal plasma or physiological NaCl solution will be prepared according to a prearranged randomization list by a technician.

The success rate will be the number of diagnosed pregnancies and live births.

DETAILED DESCRIPTION:
All couples planned for IVF will be asked to participate. After information and received informed consent they will be randomized into two groups.

At the time for ovum pick up during an IVF procedure either half of the amount of seminal plasma or the same amount of physiological NaCl solution will be installed around the external cervical opening in vagina.

Normally we do not use the seminal plasma but now half of it will be installed and the other half analysed regarding a number of cytokines possibly involved in the immunological preparation of the female internal genitalia.

The syringe with seminal plasma or physiological NaCl solution will be prepared according to a prearranged randomization list by a technician.

ELIGIBILITY:
Inclusion criteria:

* subjects have given informed consent
* infertility for at least 1 year
* the couple wishing IVF
* subjects aged between 20 - 40 years

Exclusion criterion:

* azoospermia

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1600 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2023-03 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 40 weeks
  Pregnancy as a viable fetus at ultrasonography around week 12 and delivery of baby

SECONDARY OUTCOMES:
Cytokine content | 40 weeks
  the amount of cytokines in seminal plasma used for deposition around the external cervical opening

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Nedstrand, PhD, Md, Principal Investigator — Ostergotland County Council, Sweden
Locations (1):
- University Hospital, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liffner S, Bladh M, Rodriguez-Martinez H, Sydsjo G, Zalavary S, Nedstrand E. Intravaginal exposure to seminal plasma after ovum pick-up does not increase live birth rates after in vitro fertilization or intracytoplasmic sperm injection treatment: a double-blind, placebo-controlled randomized trial. Fertil Steril. 2024 Jul;122(1):131-139. doi: 10.1016/j.fertnstert.2024.02.002. Epub 2024 Feb 9. PMID 38342372